CLINICAL TRIAL: NCT02414516
Title: A Phase 1a Dose-Escalation Study of OBP-801 in Patients With Advanced Solid Tumors
Brief Title: A Dose-Escalation Study of OBP-801 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oncolys BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBP-801-001
Record Dates: First submitted 2015-03-23; First posted 2015-04-10 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Solid Tumor
Keywords: HDAC; Epigenetic; Histone; Acetylation
MeSH Terms: interventions — YM753 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OBP-801 (Experimental)
  Interventions: Drug: OBP-801

INTERVENTIONS:
Drug: OBP-801 — OBP-801 will be administered IV

SUMMARY:
This Phase 1a, single center, open-label, repeat dose study will evaluate the safety, efficacy, and Pharmacokinetics of ascending doses of OBP-801 in patients with advanced solid tumors.

ELIGIBILITY:
Patient Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Histologically or cytologically confirmed metastatic or unresectable solid tumor.
* Has failed treatment with all standard therapies for their malignancy.
* Adequate Karnofsky Performance Status.
* An expected survival of at least 3 months.
* Adequate organ and bone marrow function.
* Signed informed consent form for study participation prior to screening.

Patient Exclusion Criteria

Patients presenting with any of the following will be excluded in the study:

* Clinically significant disease as defined by the protocol.
* Surgical therapy or other therapies within period as defined by the protocol.
* Any condition that will interfere with compliance with the protocol as determined by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03; Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 6 weeks

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile; AUC, Cmax, and t1/2 | 4 weeks
Objective Response (OR) | 22 weeks
Durability of Objective Response (DOR) | 22 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Heath EI, Weise A, Vaishampayan U, Danforth D, Ungerleider RS, Urata Y. Phase Ia dose escalation study of OBP-801, a cyclic depsipeptide class I histone deacetylase inhibitor, in patients with advanced solid tumors. Invest New Drugs. 2022 Apr;40(2):300-307. doi: 10.1007/s10637-021-01180-9. Epub 2021 Oct 6. PMID 34613570